CLINICAL TRIAL: NCT05325567
Title: Comparative Study of Post-Operative Outcomes of the Two-Incision Carpal Tunnel Release vs Mini-Open Carpal Tunnel Release
Brief Title: Comparative Study of Two Incision vs. Mini Open Carpal Tunnel Release
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study was not renewed.
Sponsor: University of Louisville (Other)
Collaborators: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21.0802
Record Dates: First submitted 2022-03-28; First posted 2022-04-13 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: On the day of surgery, all enrolled patients who happen to be in the list in an odd number will undergo 1 incision technique while those on the list who are in an even number will undergo 2 incision technique.
Who Masked: Investigator
Masking Description: Patients will be scheduled and added to the operative list of the day by the PI's primary nurse. The primary nurse is not a part of the study and will not be present in the operating room. On the day of surgery, all enrolled patients who happen to be in the list in an odd number will undergo 1 incision technique while those on the list who are in an even number will undergo 2 incision technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 incision technique (Active Comparator): a mini-open incision that allows adequate exposure of the transverse carpal ligament (TCL), while staying distal to the distal wrist crease.
  Interventions: Procedure: Mini open incision CTR
- Two incision technique (Active Comparator): A two-incision open carpal tunnel release techniques to ensure complete release both proximally and distally
  Interventions: Procedure: Mini open incision CTR

INTERVENTIONS:
Procedure: Mini open incision CTR — two techniques commonly used for carpal tunnel release are being compared to determine if one vs. the other provides superior patient outcomes.
  Other Names: Two incision CTR

SUMMARY:
Hand surgeons have many options to perform carpal tunnel release surgery. Some surgeons believe that techniques are best kept simple: a mini-open incision that allows adequate exposure of the transverse carpal ligament (TCL), while staying distal to the distal wrist crease will offer good outcomes. Others feel that as a minimally invasive technique, it is integral to spare the soft tissue structures superficial to the TCL.

This study aims to determine whether sparing these superficial structures indeed improves patient outcomes, compared to a conventional two incision approach.

DETAILED DESCRIPTION:
Carpal tunnel release (CTR) is a common surgery done by hand surgeons. The aim of the procedure is to decompress the median nerve at the level of the wrist and alleviate patient symptoms that include numbness, pain and tingling sensations along the median nerve distribution. Many versions of the technique have been described, with each description claiming improvement of post-operative results and decreasing complications.

The first description of carpal tunnel release is believed to be that of Learmonth in 1933 where he describes incising the transverse carpal ligament in a lady with a wrist fracture1. Since then, the understanding towards carpal tunnel syndrome has markedly improved, and various surgical techniques have been developed.

Because carpal tunnel syndrome has become such a common condition among the population, much knowledge has been gained about carpal tunnel surgery as well. One of the easily avoided complications of the procedure is scar related morbidity and pillar pain. Bromley offered a mini-palm open carpal tunnel release technique that decompressed the median nerve while keeping the entirety of the incision distal to the wrist crease. Tsai et al and Wilson also offered two-incision open carpal tunnel release techniques in order to keep incisions small but ensure complete release both proximally and distally. Endoscopic techniques were also eventually developed with the aim of a complete release while avoiding scar related complications.

With the many options surgeons have on how to decompress the median nerve, some begin to question if techniques are being made unnecessarily complicated. Some believe that techniques are best kept simple: a mini-open incision that allows adequate exposure of the transverse carpal ligament (TCL), while staying distal to the distal wrist crease will offer good outcomes. Others feel that as a minimally invasive technique, it is integral to spare the soft tissue structures superficial to the TCL.

This study aims to determine whether sparing these superficial structures indeed improves patient outcomes.

Hypothesis:

Null hypothesis: There is no difference in post-operative outcomes between a mini-open carpal tunnel release and a two incision carpal tunnel release

Alternative hypothesis: A two-incision carpal tunnel release will yield improvement in post operative outcomes compared to that of the mini-open carpal tunnel release

Aim of the Study:

This study aims to determine whether sparing of the soft tissue structures superficial to the transverse carpal ligament will improve post-operative outcomes of patients undergoing carpal tunnel surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants over the age of 18
* Patients who have not undergone any prior wrist surgery that may alter the native wrist anatomy
* Participants surgery must only be carpal tunnel release (no trigger fingers, de quervain release, etc.)
* Participants must have read and understood the consent form for the performance of the procedure and enrollment into the study. Consent must be signed in front of the principal investigator and a witness

Exclusion Criteria:

* Patients who are under the age of 18
* Patients who had other major surgery on the extremity being assessed potentially altering the native anatomy of the volar wrist area
* Patients who plan to have multiple hand procedures done along with their carpal tunnel release
* Patients refusing to sign the consent and enrollment form for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Resolution of carpal tunnel symptoms | Six weeks
  Reporting 2 or less on the 0-10 pain scale, with 0 as no pain

SECONDARY OUTCOMES:
Time to return to work | Six weeks
  How long it takes the subject to return to work

OTHER OUTCOMES:
2 week post operative pain | two weeks
  Reported level of pain on 0-10 pain scale, with 0 as no pain

CONTACTS AND LOCATIONS:
Overall Officials: Huey Tien, MD, Principal Investigator — University of Louisville
Locations (1):
- Kleinert Kutz Hand Care Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No